CLINICAL TRIAL: NCT05491811
Title: Evaluate the Efficacy and Safety of Ensartinib and Bevacizumab in Patients With Advanced, ALK-Rearranged Combined With TP53 Mutation, Non-Small Cell Lung Cancer: A Prospective, Open-label, Multi-center, Single-arm, Phase II Trial
Brief Title: Ensartinib in Combination With Bevacizumab in ALK-positive NSCLC Patients With TP53 Mutation
Acronym: EAGLE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Shenyang Chest Hospital (Other); Hebei Medical University Fourth Hospital (Other); First People's Hospital of Foshan (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou Institute of Respiratory Disease (Other); Central People's Hospital of Zhanjiang (Other); Guangdong Provincial Agricultural Reclamation Central Hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); West China Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Yuebei People's Hospital (Other); Yunnan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-EN-IV010
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ensartinib and Bevacizumab (Experimental): Ensartinib 225 mg oral once daily with Bevacizumab 7.5mg/kg intravenous every 3 weeks
  Interventions: Drug: Ensartinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Ensartinib — Participants will receive Ensartinib 225 mg oral once daily from baseline until disease progression, unacceptable toxicity, withdrawal of consent or death.
Drug: Bevacizumab — Participants will receive 7.5 mg/kg intravenous on Day 1 of 21 day cycles (every 3 weeks) from baseline until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Other Names: MIL60

SUMMARY:
This is a prospective, single-arm, multicenter, phase II study to investigate the efficacy and safety of Ensartinib plus Bevacizumab in metastatic anaplastic lymphoma kinase (ALK)-rearranged Non-Small Cell Lung Cancer (NSCLC) with TP53 mutation.

DETAILED DESCRIPTION:
Patients with advanced or metastatic NSCLC with ALK positive and TP53 mutation were clinically confirmed. Medical history collection, physical examination, laboratory examination, concomitant diseases and medication records were taken according to the patient's diagnosis and treatment. Laboratory examination included but not limited to blood routine and blood biochemical examination. To determine whether patients were suitable for treatment with Ensartinib combined with Bevacizumab according to the entry and exclusion criteria. For patients who met the prescription, blood samples were collected within 1 week before medication. Imaging examination was performed every 6 weeks (±7 days) in the first 2 years and every 12 weeks (±7 days) in the second 2 years. Examination items included chest CT, head MRI; See if additional tests (e.g., bone scan, total abdominal augmentation) are needed based on the actual clinical situation. When the disease progresses, blood samples should be collected within 4 weeks after the disease progression, and if possible, tumor tissues of the progressive lesions after the disease progression should be collected. Patients can choose to continue to use the regimen recommended by the doctor if the doctor considers that the use of Ensartinib therapy or combination therapy may still bring benefit to the patient. The follow-up treatment plan, the best efficacy evaluation, and the duration of treatment were recorded. When the end point of follow-up was reached, that is, the patient died or was lost to follow-up, the date of death or loss and the main causes should be tracked and recorded in detail.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced (stage IIIB) or metastatic (stage IV) NSCLC;
* ALK positive with TP53 mutation was confirmed by tissue samples or blood in each center; TP53 mutation detection needs to be confirmed by NGS. ALK positive can be detected by NGS,IHC,RT-PCR and FISH;
* Age ≥ 18 years old;
* ALK-TKI-naive patients, and allowed to have received at most one line previous chemotherapy;
* ECOG Performance status (PS) score is 0-2;
* Karnofsky Performance Status of ≥70;
* Subjects with CNS metastases are only eligible if the CNS metastases are adequately treated with radiotherapy and/or surgery and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 1 week prior to randomization.

A.Patients receiving radiotherapy or radiosurgery with a dose exceeding 30 Gy will have 3 weeks for neurological stabilization before randomization.

B.This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.

* Life expectancy of at least 12 weeks;
* Able to swallow oral drugs;
* It has certain organ system functions, defined as follows:

A. Absolute neutrophil count (ANC) ≥1.5 x 109/L B. Platelets ≥100 x 109/L C. hemoglobin ≥9 g per deciliter (≥90g per liter) note that blood transfusions are permitted to achieve the required hemoglobin level.

D. Total bilirubin ≤1.5 times upper limit of normal (ULN) E. In the absence of liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; In case of liver metastasis, ≤5×ULN.

F. Creatinine ≤1.5 x ULN. If ≥ 1.5 × ULN and creatinine clearance value calculated by Cockcroft-Gault method ≥ 50 mL/min (0.83 mL/s), patients were still eligible for inclusion.

* Female subjects of reproductive age must undergo a negative serum pregnancy test within 3 days before the start of the study medication and be willing to use a medically approved highly effective contraceptive measure (e.g., intrauterine device, contraceptive pill, or condom) during the study and within 3 months after the last administration of the study medication; Male subjects with a female partner of reproductive age should be surgically sterilized or agree to use an effective method of contraception during the study period and for 3 months after the last study dose.
* Willing and able to follow the test and follow-up procedures.
* Be able to understand the nature of the trial and complete the signing of written informed consent.

Exclusion Criteria:

* Only ALK positive or TP53 mutation;
* Patients who have received any previous ALK-TKI treatment;
* Subjects with known EGFR mutations which are sensitive to available targeted inhibitor therapy (including, but not limited to, deletions in exon 19 and exon 21 [L858R] substitution mutations) are excluded. All subjects with non-squamous histology must have been tested locally for EGFR mutation status; use of an FDA-approved test is strongly encouraged (EGFR mutation testing may be performed during the Screening Period, Non-squamous subjects with unknown or indeterminate EGFR status may not be included);
* Subjects with untreated CNS metastases are excluded;
* Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period;
* Active hepatitis B (serum HBV DNA≥1.0E+4 copies /ml[i.e. 2,000 IU/ml]), positive for hepatitis C virus antibody, HIV antibody, and treponema pallidum antibody;
* Women of childbearing age who had a positive serum pregnancy test 7 days before the start of treatment, women who were pregnant or lactating, or male and female subjects who did not take effective contraceptive measures or planned to have children during the whole treatment period and 3 months after the end of treatment;
* Patients who have used any of the following drugs within 14 days before the first dose or need to combine them during treatment: drugs at risk for prolonged QTc and/or torsive-tip ventricular tachycardia; CYP3A strong inhibitor or strong inducer;
* Major surgery or immunotherapy was performed within 4 weeks before the first dose; He received radiotherapy within 2 weeks before the first dose.
* Imaging (CT or MRI) showed that the tumor invaded the great blood vessels or it was judged that the tumor was very likely to invade the important blood vessels and cause fatal massive bleeding during the subsequent study
* Previous interstitial lung disease, drug-induced interstitial disease, or any clinically documented active interstitial lung disease; CT scan at baseline revealed the presence of idiopathic pulmonary fibrosis
* Other severe, acute, or chronic medical conditions, including uncontrolled diabetes or medical or psychiatric disorders or laboratory abnormalities, that, in the opinion of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of the study results;
* Other circumstances deemed inappropriate by the investigator for participation in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
12-month Progression-free Survival (PFS) rate | The primary analysis of 12-month PFS rate based on investigator assessment will occur when PFS maturity is observed at approximately 12 months after the first patient begin study treatment
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Progression-free survival (PFS) is defined as the time from beginning of study treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable Response Evaluation Criteria in Solid Tumors (RECIST) assessment.

SECONDARY OUTCOMES:
PFS | Through study completion, an average of 18 months
  PFS using Investigator assessment as defined by RECIST 1.1. PFS is defined as the time from beginning of study treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy prior to progression. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
Objective Response Rate (ORR) | 8 weeks
  ORR was defined as the percentage of participants who attained Complete Response (CR) or Partial Response (PR). As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Duration of Response (DoR) | 12 months
  DOR was defined as the time from when response (CR or PR) was first documented to first documented disease progression or death
Disease Control Rate (DCR) | through study completion, an average of 12 months
  DCR was defined as the proportion of CR+PR+SD subjects to total subjects
Overall Survival (OS) | Through study completion, an average of 18 months
  OS was defined as the time from randomization to death from any cause.
Disease-related symptom improvement | 12 weeks since treatment start
  To measure disease-related symptoms we will apply the Lung Cancer Symptom Scale (LCSS). The LCSS is designed as a disease-specific measure of quality of life particularly for use in clinical trials. It evaluates six major symptoms associated with lung malignancies and their effect on overall symptomatic distress, functional activities, and global quality of life. The scale consists of two segments, one completed by the patient (9 items) and one completed by the health care professional (6 items). Scoring is assigned as follows: The patient scale consists of 9 visual analogue scales (100 mm horizontal line). Patient puts a mark on line to indicate intensity of response to the items in question (0 = lowest rating). The observer scale consists of a 5-point categorical scale (100=none; 75=mild; 50=moderate; 25=marked; 0=severe). The score is equal to the length of line marked by patient. An average of the aggregate score of all 9 items is the total score (0-100, 0= least symptom burden).

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Li, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No